CLINICAL TRIAL: NCT05550818
Title: Influence of Ultra-processed Foods on Reward Processing and Energy Intake
Brief Title: Young Adult Eating Habits
Acronym: YAEH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Alexandra DiFeliceantonio, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 22-253
Record Dates: First submitted 2022-09-09; First posted 2022-09-22 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Eating Behavior; Eating Habit
Keywords: Ultra-processed food; Minimally-processed food; Executive Functioning; Eating Habits; Reward Sensitivity; Brain Activity; fMRI
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be blind to what diet is being provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Ultra Processed Food Diet (Experimental): Participants will consume a diet containing 81% total energy from UPF for 2 weeks.
  Interventions: Other: High Ultra Processed Food Diet
- No Ultra Processed Food Diet (Experimental): Participants will consume a diet containing 0% total energy from UPF for 2 weeks.
  Interventions: Other: No Ultra Processed Food Diet

INTERVENTIONS:
Other: High Ultra Processed Food Diet — Participants will be provided and consume a diet emphasizing UPF (81% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Arms: High Ultra Processed Food Diet
Other: No Ultra Processed Food Diet — Participants will be provided and consume a diet containing no UPF (0% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Arms: No Ultra Processed Food Diet

SUMMARY:
Most individuals with obesity become so before age 35 and adolescent's unhealthy dietary patterns, specifically high intake of ultra-processed foods and poor overall diet quality, may contribute to energy overconsumption and weight gain. The overall objective of this research is to establish proof-of-concept for altered reward processing measured by brain response to ultra-processed foods, an increase in ad libitum energy intake, and adverse effects on executive function in response to an ultra-processed diet (81% total energy) compared to a diet emphasizing minimally processed foods in individuals aged 18-25 years.

DETAILED DESCRIPTION:
Most individuals with obesity become so before age 35. In the US population, adolescents have the highest ultra- processed food consumption (68% of total energy) and the lowest diet quality. Given that ultra-processed foods represent two-thirds of the energy consumed by adolescents and young adults, research is needed to understand the influence of food processing on eating behaviors, particularly in the late adolescence and early adulthood life stage. During this time, individuals have increasing independence in food choice and it represents a key developmental period for executive function, processes that affect life-long mental and physical health. Evidence from pre-clinical studies demonstrates rodents maintained on a "cafeteria diet" comprised of ultra- processed ingredients have greater energy intake, weight gain, and alterations in brain circuitry that regulates both energy intake and executive function than those exposed to a standard diet. However, the impact of ultra- processed foods on the brain circuits underlying reward processing, food intake regulation, food choice, and executive function in humans is unknown. Controlled diet interventions are needed to fill this void. The overall objective of this research is to establish proof-of-concept for altered reward processing measured by brain response to an ultra-processed milkshake, an increase in ad libitum energy intake in a buffet meal, and adverse effects on executive function in response to a diet high in ultra-processed foods (81% total energy) compared to a diet emphasizing un/minimally-processed foods in individuals aged 18-25 years. To address our objective, 32 individuals aged 18-25 years (late adolescence/early adulthood) (BMI<30) will undergo two 14-day controlled feeding conditions in a randomly assigned order. Diets will match the caloric needs of the individual and be matched for potential confounding factors including macronutrients, fiber, and energy density. To assess changes in reward processing, brain response to an ultra-processed milkshake will be assessed via functional magnetic resonance imaging before and after each feeding period (4 measurements). Measurements immediately following each feeding period will include ad libitum energy intake and food selection at a breakfast buffet meal (containing both ultra-processed and minimally processed foods), eating in the absence of hunger post-meal, and executive function. Although consumption of ultra-processed foods may contribute to dysregulation of energy intake, mechanisms are uncertain and existing dietary guidelines do not address ultra- processed food intake due to a lack of human experimental research. The proposed research could address this gap and inform dietary guidelines for individuals at a critical developmental life stage - late adolescence to early adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 years
* Weight stable (+5 lbs) for previous 6 months
* No plans to gain/lose weight or change physical activity level
* Willing to pick up food daily and consume foods provided for two 14-day periods
* Verbal and written informed consent
* Unrestrained eater (TFEQ cognitive restraint score <11)
* No reported history of eating disorders
* Sedentary to recreationally active
* ADHD medications if same med >3 months at time of study

Exclusion Criteria:

* BMI >30 kg/m2
* Endocrine disorders or other major chronic disease (e.g., type 2 diabetes, hypothyroidism, hypertension)
* Pregnant or plans to become pregnant
* Food allergies or aversions
* Claustrophobia
* History of head injury with loss of consciousness for more than 10 minutes
* Contraindications to MRI: individuals with pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra G DiFeliceantonio, PhD, Principal Investigator — Virginia Polytechnic Institute and State University; Brenda M Davy, PhD, RDN, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - Virginia Polytechnic Institute and State University, Blacksburg, Virginia
  - Fralin Biomedical Research Institute at VTC, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rego MLM, Leslie E, Schmall E, Capra B, Hudson S, Ahrens ML, Katz B, Davy KP, Hedrick VE, DiFeliceantonio AG, Davy BM. The Influence of Ultraprocessed Food Consumption on Energy Intake in Emerging Adulthood: A Controlled Feeding Trial. Obesity (Silver Spring). 2025 Nov 19. doi: 10.1002/oby.70086. Online ahead of print. PMID 41255123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 individuals were screened for eligibility between March 10, 2023 and September 1, 2024 in Blacksburg, VA.
Pre-assignment Details: 33 of 36 participants were randomized. Of those not randomized, 1 did not meet inclusion criteria, 1 was lost to follow up, and 1 voluntarily withdrew due to time commitment.
Groups:
- High Ultra Processed Food Diet First, Then No Ultra Processed Food Diet: Participants will consume a diet containing 81% total energy from UPF for 2 weeks.
  High Ultra Processed Food Diet: Participants will be provided and consume a diet emphasizing UPF (81% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 0% total energy from UPF for 2 weeks.
- No Ultra Processed Food Diet First, Then Ultra Processed Food Diet: Participants will consume a diet containing 0% total energy from UPF for 2 weeks.
  No Ultra Processed Food Diet: Participants will be provided and consume a diet containing no UPF (0% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 81% total energy from UPF for 2 weeks.
Period: Overall Study
Arm/Group | High Ultra Processed Food Diet First, Then No Ultra Processed Food Diet | No Ultra Processed Food Diet First, Then Ultra Processed Food Diet
Started | 15 | 18
Completed | 12 | 16
Not Completed | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Ultra Processed Food Diet First: Participants will consume a diet containing 81% total energy from UPF for 2 weeks.
  High Ultra Processed Food Diet: Participants will be provided and consume a diet emphasizing UPF (81% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 0% total energy from UPF for 2 weeks.
- No Ultra Processed Food Diet First: Participants will consume a diet containing 0% total energy from UPF for 2 weeks.
  No Ultra Processed Food Diet: Participants will be provided and consume a diet containing no UPF (0% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 81% total energy from UPF for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | High Ultra Processed Food Diet First | No Ultra Processed Food Diet First | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.73 (2.15) | 22.00 (1.97) | 21.88 (2.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 1
  Asian or Pacific Islander | 2 | 4 | 6
  Black or African American | 0 | 0 | 0
  White | 10 | 13 | 23
  Other | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Response From Baseline to 2-weeks Post High UPF or 2 Weeks no UPF Diet
Description: Brain response to milkshake was measured using functional magnetic resonance imaging (fMRI). On the first level a contrast of milkshake > tasteless was built. The measures presented here are the beta values of the milkshake>tasteless contrast extracted from an orbital frontal cortex apriori region of interest. The pre intervention beta values were subtracted from the post intervention values. Extracted beta values are by definition arbitrary units and are the standard measure for fMRI.
Time Frame: 4 measurements (pre/post 2-week UPF diet, pre/ post 2-week no UPF diet)
Population: Of the 28 participants that completed the study, 24 were analyzed. Data collection was not completed for one participant due to a power outage. 2 participants were excluded due to excess motion in the scanner. 1 participant was ill at the time of assessment.
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- High Ultra Processed Food Diet: Participants will consume a diet containing 81% total energy from UPF for 2 weeks.
  High Ultra Processed Food Diet: Participants will be provided and consume a diet emphasizing UPF (81% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 0% total energy from UPF for 2 weeks.
- No Ultra Processed Food Diet: Participants will consume a diet containing 0% total energy from UPF for 2 weeks.
  No Ultra Processed Food Diet: Participants will be provided and consume a diet containing no UPF (0% energy). Diets will be eucaloric (50% carbohydrate, 35% fat,15% protein) matched for dietary soluble and insoluble fiber, added sugar, mono- and polyunsaturated fat, saturated fat, antioxidant nutrients, sodium, and overall diet quality, for 2 weeks.
  Next, participants will consume a diet containing 81% total energy from UPF for 2 weeks.
Arm/Group | High Ultra Processed Food Diet | No Ultra Processed Food Diet
Number analyzed (Participants) | 24 | 24
arbitrary units | 0.02 (0.51) | 0.13 (0.76)

2. Secondary Outcome: Change in Energy Intake From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: Participants will arrive at the laboratory in the fasted state for an ad libitum breakfast buffet meal. The buffet meal will contain a variety of food items that vary in macronutrient content and in their degree of processing (UPF, no UPF). The meal will consist of typical breakfast items in excess of what would normally be consumed. Participants will self-select foods over a 30-minute period. Food items will be weighed (±0.1 grams) prior to and after the completion of the meal to determine the amount consumed (g, kcal), calculated using NDSR nutritional analysis software.
Time Frame: 2 measurements following the 2-week UPF diet (day 15), following the 2-week no UPF diet (day 15)
Reporting Status: Not Posted

3. Secondary Outcome: Change in Eating Rate From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: Participants will arrive at the laboratory in the fasted state for an ad libitum breakfast buffet meal. The buffet meal will contain a variety of food items that vary in macronutrient content and in their degree of processing (UPF, no UPF). The meal will consist of typical breakfast items in excess of what would normally be consumed. Participants will self-select foods over a 30-minute period. Meal eating rate (g/min, kcal/min) will be determined using meal start and stop times.
Time Frame: 2 measurements following the 2-week UPF diet (day 15), following the 2-week no UPF diet (day 15)
Reporting Status: Not Posted

4. Secondary Outcome: Change in Food Items Selected From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: At the ad libitum buffet meal, food selection will be determined by the number of items consumed from UPF vs no UPF.
Time Frame: 2 measurements (following the 2-week UPF diet, following the 2-week no UPF diet)
Reporting Status: Not Posted

5. Secondary Outcome: Change in Grams of Food Selected From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: At the ad libitum buffet meal, food selection will be determined by the number of grams consumed from UPF vs no UPF.
Time Frame: 2 measurements (following the 2-week UPF diet, following the 2-week no UPF diet)
Reporting Status: Not Posted

6. Secondary Outcome: Change in Amount of Energy (Kcals) Selected From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: At the ad libitum buffet meal, food selection will be determined by the number of amount of energy (kcals) consumed from UPF vs no UPF.
Time Frame: 2 measurements (following the 2-week UPF diet, following the 2-week no UPF diet)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Executive Function From Baseline to 2-weeks Post High UPF or 2 Weeks no UPF Diet
Description: Participants will undergo computerized tests of executive function, such as working memory, cognitive flexibility, and inhibitory control. These tasks have been widely used with participants across the lifespan and contain simple graphics.
Time Frame: 4 measurements (pre/post 2-week UPF diet, pre/ post 2-week no UPF diet)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Eating in the Absence of Hunger From Baseline to 2-weeks Post High UPF or 2 Weeks no UPF Diet
Description: Following the ad libitum buffet meal, participants will move to a separate room where an ample amount of 4 pre-weighed snack items (2 UPF, 2 no UPF) and magazines are available. Using an approach consistent with previous research studying this outcome, participants will be instructed to take 2 bites of each snack item and rate its palatability on the LHS, and to eat the remainder of the snacks or look at the magazines while they wait for the next part of the study. Participants will be left to consume the snacks or relax for 15 minutes. Participants will also be given a box of snacks to assess eating in the absence of hunger outside the laboratory environment. Snack boxes will be returned to study staff the next morning. Staff will document the amount and type of snacks consumed.
Time Frame: 4 measurements (in person and take home portion following the 2-week UPF diet, in person and take home portion following the 2-week no UPF diet)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Internal State Ratings From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: To assess sensations of hunger a Visual Analog Scale bounded by "not hungry at all" and "extremely hungry" will be used. With higher scores indicated higher hunger. Same for fullness. Visual Analog Scales will be completed prior to (min. 0), and following the buffet meal (min. 30).
Time Frame: 2 measurements (following the 2-week UPF diet, following the 2-week no UPF diet)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Sensitivity to Delayed Consequences From 2 Weeks High UPF or 2 Weeks no UPF Diet
Description: To assess sensitivity to delayed consequences by assessing preference for different amounts of money varying over different amounts of time. This will be associated with a k value (discount rate), the lower the k value, the less discounting.
Time Frame: 4 measurements (pre/post 2-week UPF diet, pre/ post 2-week no UPF diet)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 21 months
Arm/Group | High Ultra Processed Food Diet First | No Ultra Processed Food Diet First
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT05550818/Prot_SAP_000.pdf